CLINICAL TRIAL: NCT02859519
Title: A Multi-centre, Double-blind, Randomized, Vehicle-controlled Study of Efficacy and Safety of Topical MOB015B in the Treatment of Mild to Moderate Distal Subungual Onychomycosis (DSO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOB015B-IV
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Distal Subungual Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- MOB015B (Experimental): Subjects will treat all affected fingernails and/or toenails with MOB015B for 48 weeks once daily at bedtime.
  Interventions: Drug: MOB015B
- MOB015B Vehicle (Placebo Comparator): Subjects will treat all affected fingernails and/or toenails with MOB015B Vehicle for 48 weeks once daily at bedtime.
  Interventions: Drug: MOB015B Vehicle

INTERVENTIONS:
Drug: MOB015B — MOB015B - Terbinafine hydrochloride (HCl) 10%, topical solution
  Arms: MOB015B
Drug: MOB015B Vehicle — MOB015B Vehicle without the active ingredient Terbinafine
  Arms: MOB015B Vehicle

SUMMARY:
The primary objective of this study is to evaluate the efficacy of topical MOB015B in patients with mild to moderate distal subungual onychomycosis (DSO).

The secondary objective is to evaluate the safety of topical MOB015B in patients with mild to moderate DSO.

DETAILED DESCRIPTION:
Male or female subjects aged between 12 and 75 years with confirmed DSO involving 20-60% of at least one great toenail will be screened for randomization in this study. The diagnosis of DSO will be confirmed prior to randomization through a positive culture of dermatophytes. In addition, a central blinded assessment of the clinical disease involvement (i.e., affected nail area) will be performed at Screening. Subjects have to meet all eligibility criteria before being randomized in to the study.

Eligible subjects will be randomized to the investigational medicinal products (MOB015B or vehicle) in a ratio of 2:1. The investigational medicinal products (IMPs) will be applied to all affected fingernails and/or toenails for 48 weeks once daily at bedtime. However, fingernails will not be assessed for efficacy.

Since both the IMPs are indistinguishable in appearance and mode of administration, the study will be performed as a double-blind study, i.e., both the investigator and the subject will remain blinded throughout the entire study.

After a 4-week follow-up period without IMP treatment the end of study (EoS) Visit will be performed at Week 52 (Visit 7). The primary efficacy variable will be assessed at Week 52. The end of the clinical study for each individual subject is defined as the EoS Visit at Week 52 (Visit 7). The end of the clinical study is defined as the last visit of the last subject in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 12 - 75 years of age
2. Distal subungual onychomycosis (DSO) of at least one of the great toenail(s) affecting 20% to 60% of the target nail
3. Positive culture for dermatophytes
4. Written informed consent

Exclusion Criteria:

1. Proximal subungual onychomycosis
2. Distal subungual onychomycosis of both great toenails where involvement has extended into the proximal portion of the target nail (unaffected proximal nail is less than 3 mm)
3. Target toenail thickness more than 3 mm
4. "Spike" of onychomycosis extending to eponychium of the target toenail
5. Presence of dermatophytoma (defined as thick masses of fungal hyphae and necrotic keratin between the nail plate and nail bed) on the target nail
6. Other conditions than DSO known to cause abnormal nail appearance
7. Presence of toenail infection other than dermatophytes
8. Previous target toenail surgery with any residual disfigurement
9. Topical treatment of the nails with other antifungal medication within 6 weeks before screening/Visit 1
10. Systemic use of antifungal treatment within 6 months before screening/visit 1
11. Severe moccasin tinea pedis
12. Signs of severe peripheral circulatory insufficiency
13. Uncontrolled diabetes mellitus
14. Known immunodeficiency
15. Participation in another clinical trial with an investigational drug or device during the previous 3 months before Baseline/ Visit 2
16. Known allergy to any of the tested treatment products
17. A positive pregnancy test at Baseline/Visit 2 indicating pregnancy in a woman of childbearing potential or a premenarche subject
18. Females who are pregnant or breastfeeding
19. Men who have female sexual partners of child-bearing potential and sexually active women of child-bearing potential who are not practicing an acceptable method of birth control, or who will not remain abstinent through the trial.
20. Patients previously randomized in this study
21. History of, or current drug or alcohol abuse
22. Psychiatric condition that might limit the participation in the study and/or that lead to the assumption that the patient's ability to completely understand the consequences of consent is missing
23. Close affiliation with the investigator (e.g. a close relative) or persons working at a study site, or patient who is an employee of the sponsor's company
24. Patients who are institutionalized because of legal or regulatory order
25. Any diseases or circumstances in which the patient should not participate in the study in the opinion of the investigator

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Subjects with complete cure of the target toe nail at Week 52 | Week 52
  Complete cure was defined as negative fungal culture of dermatophytes, negative direct potassium hydroxide (KOH) microscopy and 0% clinical disease involvement of the target toenail.

SECONDARY OUTCOMES:
Subjects with mycological cure of the target toe nail at Week 52 | Week 52
  Mycological cure was defined as negative fungal culture of dermatophytes and negative direct KOH microscopy of the target toenail.
Subjects with treatment success of the target toe nail at Week 52 | Week 52
  Treatment success was defined as negative fungal culture of dermatophytes, negative direct KOH microscopy and ≤10% clinical disease involvement of the target toenail.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - Multiple Locations, California
  - Multiple Locations, Florida
  - Multiple Locations, Idaho
  - Rolling Meadows, Illinois
  - Fridley, Minnesota
  - Multiple Locations, New Jersey
  - Multiple Locations, Oregon
  - Multiple Locations, Texas
  - Multiple Locations, Virginia
- Multiple Locations, Canada